CLINICAL TRIAL: NCT04231734
Title: Pilot Phase I Study of Ketogenic Diet in the Treatment of Patients With Untreated Mantle Cell Lymphoma With a Low Tumor Burden
Brief Title: Ketogenic Diet in Patients With Untreated Low Tumor Burden Mantle Cell Lymphoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-05020213
Record Dates: First submitted 2019-12-30; First posted 2020-01-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Mantle Cell Lymphoma; Ketogenic Dieting
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Low tumor burden, treatment-naïve MCL
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — Prepared ketogenic meals, 3 per day for up to 12 weeks (Day 1 through Day 84)

SUMMARY:
This study evaluates adherence to a ketogenic diet in patients with low tumor burden, treatment-naïve mantle cell lymphoma.

DETAILED DESCRIPTION:
This is a single-arm feasibility study to evaluate adherence to a ketogenic diet in patients with low tumor burden, treatment-naïve mantle cell lymphoma.

Subjects will be evaluated for eligibility and baseline assessments prior to initiating the ketogenic diet during the screening period and/or prior to initiating the ketogenic diet on Day 1. Eligible subjects will receive study treatment which will consist of a daily ketogenic diet for up to 12 weeks (Day 1 through Day 84). Subjects will be monitored with weekly assessments of adherence to diet and effects on serum metabolic markers, tumor specimens, and body composition.

After discontinuing the ketogenic diet, subjects will be followed for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of mantle cell lymphoma
* Age ≥ 18 years
* No prior systemic therapy for lymphoma
* ECOG performance status ≤ 2
* Required initial laboratory parameters:

  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
  * Platelet count ≥ 75,000 cells/mm3
  * Calculated creatinine clearance ≥ 30 ml/min by Cockcroft-Gault formula
  * Total bilirubin ≤ 2.0 x ULN
  * AST/SGOT or ALT/SGPT ≤ 3.0 x ULN
* Understand and voluntarily sign an ICF prior to any study related assessments and procedures are conducted

Exclusion Criteria:

* Patients with blastoid histology
* Patients with known or suspected central nervous system (CNS) involvement
* Patients with a clear indication for treatment of lymphoma, including those with a tumor larger than 6 cm, more than 3 lymph nodes more than 3 cm, or constitutional symptoms
* Active viral infection with HIV or hepatitis type B or C. Seropositive HBV patients are eligible if they are negative for HBV DNA by PCR and receive concomitant antiviral therapy during treatment and for additional six months after coming off study.
* Active uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* Uncontrolled moderate to severe hypertriglyceridemia (TG>300 mg/dL).
* Strong family history of hypertriglyceridemia and coronary artery disease.
* Myocardial infarction within 6 months of cycle 1, day 1. [Subjects with a history of myocardial infarction between 6 and 12 months prior to cycle 1, day 1, who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event, may participate].
* Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV. In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥ 2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction < 40% by multigated acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI).
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication.
* Patients requiring dual anti-platelets treatment for cardiac conditions or patients who are on anticoagulation for arterial or venous thrombosis.
* Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Type I diabetes
* Uncontrolled Type II diabetes mellitus (HbA1c> 7.5%).
* Type II diabetes requiring treatment with a sulfonylurea, meglitinide, or insulin.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Active complaints of dysphagia or odynophagia
* Presence of a "feeding tube" (i.e. nasogastric tube, PEG, PEJ)
* Participation in a specialty diet (e.g. Atkins, Weight Watchers, Best Life, Nutrisystem, South Beach, Jenny Craig, Paleo Diet, Zone, etc) or weight loss plan within 28 days prior to Cycle 1 of treatment.
* Vegetarian or vegan eating habits.
* An allergy or intolerance to egg, gluten, tree nuts, or milk protein.
* History of serious or uncontrolled gout or hyperuricemia
* Diagnosis of a seizure disorder.
* Prior diagnosis of restless legs syndrome or a history of chronic muscle cramps, as defined as a period of at least 1 month where spontaneous cramping of the skeletal muscles occurred more than two-thirds of the days.
* Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through at least 30 days after the last dose of trial treatment.
* History of nephrolithiasis or nephrolithiasis incidentally discovered during CT screening.
* Known selenium deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who adhere to ketogenic diet | 12 weeks
  Number of subjects who adhere to ketogenic diet as defined by serum betahydroxybutyrate > 1.0 mM at 7 out of 11 timepoints

SECONDARY OUTCOMES:
Number of subjects who achieve a partial or complete response | 12 weeks
  Number of subjects who achieve a partial or complete response based on radiographic imaging using Lugano criteria for lymphoma response
Number of subjects who exhibit a significant change in fasting serum metabolic markers | Baseline, 16 weeks
  Fasting metabolic markers to be assessed for this outcome measure include insulin, glucose, and lipids
Number of subjects who exhibit a significant change in serum mediators of inflammation | Baseline, 16 weeks
  Serum mediators of inflammation to be assessed for this outcome measure include high sensitivity C-reactive protein (hs-CRP), interleukin (IL)-6, tumor necrosis factor (TNF)-a, IL-1beta, and interferon (INF)-gamma.
Number of subjects who exhibit a significant change in blood cell populations | Baseline, 16 weeks
  Blood cell populations will be assessed by performance of unbiased expression analysis (RNA-Seq) from blood cell populations, and High-Dimensional Single-Cell Mass Cytometry (CyTOF) analysis of peripheral blood cells
Change in body composition as measured by difference in ideal body weight and actual body weight at the end of study compared to baseline | Baseline, 16 weeks
Number of subjects who complete quality of life questionnaires at required timepoints | 16 weeks
  Quality of life questionnaire to be used for this outcome measure is EORTC-C30
Effect of ketogenic diet on gut microbiome | 12 weeks
  Change in proportion of most common gut bacteria identified by DNA analysis of stool samples
Rate of recruitment | 1 year
  Percentage of subjects screened for the trial who eventually enroll in the trial
Subject adherence to scheduled laboratory assessments | 12 weeks
  Percentage of laboratory assessments successfully attended by subjects
Subject adherence to meal assessments | 12 weeks
  Percentage of meal assessments successfully completed by subjects
Rate of attrition | 12 weeks
  Percentage of subjects enrolled who drop out before trial completion
Rate of daily ketosis | 12 weeks
  Percentage of days in ketosis as defined by positive ketones results on ketostix

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WCM Joint Clinical Trials Office — https://jcto.weill.cornell.edu/